CLINICAL TRIAL: NCT00192335
Title: A Prospective, Double-Blind, Randomized Trial to Demonstrate Equivalent Immunogenicity of CAIV-T and FLUMIST in Healthy Participants Ages 5 Through 49 Years
Brief Title: Trial to Demonstrate Equivalent Immunogenicity of CAIV-T and FLUMIST in Healthy Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP112
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Healthy
MeSH Terms: interventions — FluMist

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): CAIVT-The total volume of 0.2 mL will be administered intranasally with a spray applicator (approximately 0.1 mL into each nostril).
  Interventions: Biological: CAIV-T; Biological: CAIVT
- 2 (Active Comparator): FluMist- The total volume of 0.5 mL will be administered intranasally with a spray applicator (approximately 0.25 mL into each nostril).
  Interventions: Biological: FluMist

INTERVENTIONS:
Biological: CAIV-T
  Arms: 1
Biological: CAIVT — The total volume of 0.2 mL will be administered intranasally with a spray applicator (approximately 0.1 mL into each nostril).
  Arms: 1
Biological: FluMist — The total volume of 0.5 mL will be administered intranasally with a spray applicator (approximately 0.25 mL into each nostril).
  Arms: 2

SUMMARY:
* Primary objective is to demonstrate equivalent immunogeniticity of CAIV-T and FluMist
* Secondary objective of this study is to assess the safety and tolerability of CAIV-T compared to FluMist

ELIGIBILITY:
Inclusion Criteria:

* Age 5 through 49 years (not yet reached their 50th birthday);
* In general good health;
* Individual or parent/guardian available by telephone;
* Ability of the participant or parent/guardian to understand and comply with the requirements of the protocol; and
* Written informed consent and HIPAA authorization obtained from the participant's parent or legal guardian or written informed consent and HIPAA authorization obtained from the participant.

Exclusion Criteria:

* History of hypersensitivity to any component of FluMist or CAIV-T, including egg or egg products;
* History of hypersensitivity to gentamicin;
* Any known immunosuppressive condition or immune deficiency disease (including HIV infection), or ongoing receipt of any immunosuppressive therapy;
* Household contact who is immunocompromised (participants should also avoid close contact with other immunocompromised individuals for at least 21 days);
* History of chronic underlying medical conditions such as chronic disorders of the cardiovascular and pulmonary systems, chronic metabolic diseases (including diabetes), renal dysfunction, or hemoglobinopathies;
* History of Guillain-Barré syndrome;
* History of asthma or reactive airways disease;
* For children age 5 through 8 years, receipt of prior influenza vaccination;
* Acute febrile (>100.0°F oral) and/or respiratory illness within the 72 hours prior to enrollment;
* For participants under the age of 18, use of aspirin or aspirin containing products in the 30 days prior to enrollment or anticipated use during the study;
* Administration of any live vaccine within 30 days prior to enrollment or if receipt of another live vaccine is expected within 30 days of the vaccination in this study;
* Administration of any inactivated vaccine within two weeks prior to enrollment or if receipt of another inactivated vaccine is expected within two weeks of the vaccination in this study;
* Pregnancy or, in biologically capable women (e.g., menses within the last year), not willing to agree to acceptable birth control for 90 days after enrolling into the study (for those biologically capable, a urine pregnancy test must be performed on the day of vaccination with a negative result);
* Breastfeeding or lactating women;
* Participation in another investigational trial or administration of any investigational drug within 30 days prior to enrollment or during this study;
* Receipt of any blood product within 90 days prior to vaccination or expected receipt within the study duration;
* Employees of the research center, any individuals involved with the conduct of the study, or any family member of such individuals; and
* Any condition that in the opinion of the investigator would interfere with the interpretation or evaluation of the vaccine.

Ages: 5 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 890 (Actual)
Dates: Start 2004-07; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
- Among participants 5 through 8 years of age regardless of baseline serostatus who receive two doses, the post-dose two strain-specific geometric mean titers (GMTs) for serum HAI in the CAIV-T group are within 2-fold of those in the FluMist group | greater than 28-days post dose

SECONDARY OUTCOMES:
The proportion of participants experiencing each of the reactogenicity events by dose. | Within 28 days of vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Luis Angles, MD, Principal Investigator — Heart of America Research Institute
Locations (3):
- United States (3):
  - Heart of America Research Institute, Shawnee Mission, Kansas
  - Kentucky Pediatric/Adult Research, Inc., Bardstown, Kentucky
  - R/D Clinical Research, Inc., Lake Jackson, Texas